CLINICAL TRIAL: NCT01995110
Title: Identification of Nutritional Health Biomarkers for Metabolic Flexibility in Blood - a Randomized, Postprandial, Caloric Dose-response Strategy
Brief Title: Postprandial Blood Cell Transcriptome of Normal Weight and Obese Subjects to 3 Caloric Doses of a High-fat Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agroscope Liebefeld-Posieux Research Station ALP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NUTRICHIP-1-transcriptome
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Obesity; Nutritional Intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal weight subjects (Experimental)
  Interventions: Other: high-fat meal A; Other: high-fat meal B; Other: high-fat meal C
- obese subjects (Experimental)
  Interventions: Other: high-fat meal A; Other: high-fat meal B; Other: high-fat meal C

INTERVENTIONS:
Other: high-fat meal A
  Other Names: high-fat meal consisting of 500 kcal
Other: high-fat meal B
  Other Names: high-fat meal B consisting of 1000 kcal
Other: high-fat meal C
  Other Names: high-fat meal C consisting of 1500 kcal

SUMMARY:
The study will quantitatively evaluate the metabolic response of normal weight and obese subjects to three high-fat meals differing in caloric dose by analysing the postprandial blood transcriptome.

ELIGIBILITY:
Inclusion Criteria for normal weight subjects:

* age 25-50
* 20<BMI>25
* waist circumference <94cm

Inclusion Criteria for obese subjects:

* age 25-50
* 30<BMI>40
* waist circumference >102cm

Exclusion Criteria for both groups:

* physiological or psychological diseases
* allergies to food or intolerance to high-fat meal
* vegetarians, vegans
* chronic intake of drugs
* smokers
* diabetes mellitus type I and II
* debiliating kidney disease
* debiliating liver disease
* clinically established coronary heart diseases
* ingestion of vitamins or dietary supplements during the course of the study

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
blood cell transkriptome/ gene-expression | 0h, 2h, 4h, 6h
  * differently expressed genes between normal weight and obese subjects at baseline
  * changes in gene-expression 2, 4 and 6h after consumption

CONTACTS AND LOCATIONS:
Overall Officials: Guy Vergeres, PhD, Principal Investigator — Agroscope Liebefeld-Posieux Research Station ALP; Doreen Gille, M.Sc., Study Director — Agroscope Liebefeld-Posieux Research Station ALP; Kurt Laederach, MD, Study Director — Inselspital University of Berne
Locations (2):
- Switzerland (2):
  - Agroscope, Bern, Canton of Bern
  - University Hospital Inselspital Berne, Bern, Canton of Bern